CLINICAL TRIAL: NCT07129850
Title: Bempedoic Acid in Primary Percutaneous Coronary Intervention: Impact on Inflammatory Markers, Procedural and Clinical Outcomes
Brief Title: Bempedoic Acid in PPCI Impact on Clinical Outcome and Inflammatory Markers
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mostafa Sayed Ahmed, Principal Investigator, Assiut University
Other Study IDs: Bempedoic acid in PPCI
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: ST Elevation (STEMI) Myocardial Infarction
Keywords: Bempedoic acid; TNF alpha; PPCI
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Two groups will be measured

SUMMARY:
Bempedoic acid in PPCI

DETAILED DESCRIPTION:
Cardiovascular disease persists as the predominant cause of global burden of mortality and morbidity worldwide(1).

The cholesterol hypothesis posits that elevated blood cholesterol levels constitute a significant risk factor for atherosclerotic cardiovascular disease (ASCVD) and reducing cholesterol levels will consequently lower the risk of ASCVD(2).

Treatments aimed at lowering lipid levels have demonstrated their effectiveness in decelerating the advancement of atherosclerotic disease(3). This finding further reinforces the pathophysiological connections between plasma lipids and the progression of CAD. Among non-lipid mechanisms involved in reducing CAD progression, lipid-lowering drugs have also been implicated in plaque stabilization, reduced inflammation, reversal of endothelial dysfunction, and decreased thrombogenicity(3).

It is widely accepted that the beneficial effects of statins on cardiovascular events are mainly linked to their cholesterol lowering properties. Nonetheless, statins also have a clear action in reducing systemic inflammation. The effect on hsCRP is proportionally similar to that on LDL-C(4).

It is known that an anti-inflammatory action contributes to the reduction of cardiovascular risk independently of the effect on LDL-C. Four-year therapy with canakinumab, a specific anti-interleukin-1b monoclonal antibody, in patients with previous myocardial infarction reduced the relative risk of relapse by approximately 15% by reducing hsCRP levels by 60% without modifying LDL-C(5). It is therefore possible to hypothesize that cholesterol lowering drugs with an effect on hsCRP, such as statins and bempedoic acid, have advantages in reducing cardiovascular events compared to those that do not act on inflammation, such as PCSK9 inhibitors(4).

Bempedoic acid is a new cholesterol-lowering drug, which has recently received US FDA approval. It offers a safe and effective oral therapeutic option for lipid lowering in patients who cannot tolerate statins or in addition to statins in patients who are not reaching the LDL target(6). Bempedoic acid targets lipid and glucose metabolism as well as inflammation. The primary effect is the reduction of cholesterol synthesis in the liver and its administration is generally not associated to unwanted muscle effects(4).

Bempedoic acid may decrease gluconeogenesis leading to improved insulin sensitivity, glucose metabolism, and metabolic syndrome(4).

The anti-inflammatory action of bempedoic acid is mainly achieved via activation of AMPK pathway in the immune cells, leading to decreased plasma levels of C-reactive protein(4).

However, its potential role in modulating post-PCI inflammatory response has not been fully investigated, especially in primary PCI setting.

ELIGIBILITY:
Inclusion Criteria:

Age ≥18 years STEMI diagnosis Undergoing primary PCI

Exclusion Criteria:

Known allergy to Bempedoic acid Active infection or chronic inflammatory disease Severe hepatic or renal dysfunction Use of immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study Population The study will include patients presenting with ST-elevation myocardial infarction (STEMI) who are eligible for and undergoing primary percutaneous coronary intervention (PCI) at Assiut University Heart Hospital.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-08-14 (Estimated); Primary Completion 2026-08-14 (Estimated); Study Completion 2027-11-14 (Estimated)

PRIMARY OUTCOMES:
Change in inflammatory markers | At 1 month post-PCI.
  reactive protein [CRP] and tumor necrosis factor-alpha [TNF-α]) at 1 month post-primary PCI compared between the intervention group (Bempedoic Acid) and the control group.

SECONDARY OUTCOMES:
Final TIMI flow grade post-PCI. | 1 day
  Assessment of final TIMI flow grade, incidence of no-reflow phenomenon, and occurrence of contrast-induced nephropathy (CIN) after primary PCI.
Major Adverse Cardiac Events | Within 30 days post-PCI.
  Incidence of a composite endpoint including heart failure, reinfarction, rehospitalization for cardiac causes, arrhythmia, stroke, and cardiovascular mortality.
Lipid Profile Changes | At 1 month post-PCI.
  Measurement of total cholesterol, LDL-C, HDL-C, and triglycerides to assess lipid-lowering effect of Bempedoic Acid.

CONTACTS AND LOCATIONS:
Overall Officials: Amr Youssef, Professor, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Laufs U, Banach M, Mancini GBJ, Gaudet D, Bloedon LT, Sterling LR, Kelly S, Stroes ESG. Efficacy and Safety of Bempedoic Acid in Patients With Hypercholesterolemia and Statin Intolerance. J Am Heart Assoc. 2019 Apr 2;8(7):e011662. doi: 10.1161/JAHA.118.011662. PMID 30922146
- [Result] Ridker PM, Everett BM, Thuren T, MacFadyen JG, Chang WH, Ballantyne C, Fonseca F, Nicolau J, Koenig W, Anker SD, Kastelein JJP, Cornel JH, Pais P, Pella D, Genest J, Cifkova R, Lorenzatti A, Forster T, Kobalava Z, Vida-Simiti L, Flather M, Shimokawa H, Ogawa H, Dellborg M, Rossi PRF, Troquay RPT, Libby P, Glynn RJ; CANTOS Trial Group. Antiinflammatory Therapy with Canakinumab for Atherosclerotic Disease. N Engl J Med. 2017 Sep 21;377(12):1119-1131. doi: 10.1056/NEJMoa1707914. Epub 2017 Aug 27. PMID 28845751
- [Result] Biolo G, Vinci P, Mangogna A, Landolfo M, Schincariol P, Fiotti N, Mearelli F, Di Girolamo FG. Mechanism of action and therapeutic use of bempedoic acid in atherosclerosis and metabolic syndrome. Front Cardiovasc Med. 2022 Oct 28;9:1028355. doi: 10.3389/fcvm.2022.1028355. eCollection 2022. PMID 36386319
- [Result] Feingold KR. Guidelines for the Management of High Blood Cholesterol. 2025 Mar 27. In: Feingold KR, Adler RA, Ahmed SF, Anawalt B, Blackman MR, Chrousos G, Corpas E, de Herder WW, Dhatariya K, Dungan K, Hamilton E, Hofland J, Jan de Beur S, Kalra S, Kaltsas G, Kapoor N, Kim M, Koch C, Kopp P, Korbonits M, Kovacs CS, Kuohung W, Laferrere B, Levy M, McGee EA, McLachlan R, Muzumdar R, Purnell J, Rey R, Sahay R, Shah AS, Sperling MA, Stratakis CA, Trence DL, Wilson DP, editors. Endotext [Internet]. South Dartmouth (MA): MDText.com, Inc.; 2000-. Available from http://www.ncbi.nlm.nih.gov/books/NBK305897/ PMID 26247090
- [Result] WHO CVD Risk Chart Working Group. World Health Organization cardiovascular disease risk charts: revised models to estimate risk in 21 global regions. Lancet Glob Health. 2019 Oct;7(10):e1332-e1345. doi: 10.1016/S2214-109X(19)30318-3. Epub 2019 Sep 2. PMID 31488387